CLINICAL TRIAL: NCT00064246
Title: A Phase I/II Study: Zevalin Radioimmunotherapy for Patients With Post Transplant Lymphoproliferative Disease Following Solid Organ Transplantation
Brief Title: Yttrium Y 90 Ibritumomab Tiuxetan and Rituximab in Treating Patients With Post-Transplant Lymphoproliferative Disorder
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02721; AMC-037; U01CA070019 (NIH); CDR0000310158 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-07-08; First posted 2003-07-09 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: Post-transplant Lymphoproliferative Disorder; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Stage III Adult Burkitt Lymphoma; Stage III Adult Diffuse Large Cell Lymphoma; Stage IV Adult Burkitt Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Waldenström Macroglobulinemia
MeSH Terms: conditions — Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Waldenstrom Macroglobulinemia | interventions — Rituximab; Indium; ibritumomab tiuxetan

ARMS (1):
- Treatment (rituximab, yttrium Y 90 ibritumomab tiuxetan) (Experimental): Phase I: Patients receive rituximab IV and indium In 111 ibritumomab tiuxetan IV over 10 minutes on day 1. Patients undergo 2 (or 3 if needed) imaging scans between days 1-6. In the absence of altered biodistribution, patients receive rituximab IV followed within 4 hours by IDEC-Y2B8 IV over 10 minutes on day 8.
  Phase II: Patients receive treatment as in phase I at the MTD of IDEC-Y2B8. Patients are followed monthly for 3 months, every 3 months for 2 years, and then every 6 months for 2 years.
  Interventions: Biological: rituximab; Radiation: indium In 111 ibritumomab tiuxetan; Radiation: yttrium Y 90 ibritumomab tiuxetan

INTERVENTIONS:
Biological: rituximab — Given IV
  Other Names: IDEC-C2B8; IDEC-C2B8 monoclonal antibody; Mabthera; MOAB IDEC-C2B8; Rituxan
Radiation: indium In 111 ibritumomab tiuxetan — Given IV
  Other Names: IDEC-In2B8
Radiation: yttrium Y 90 ibritumomab tiuxetan — Given IV
  Other Names: 90Y ibritumomab tiuxetan; IDEC Y2B8; Y90 Zevalin; Y90-labeled ibritumomab tiuxetan

SUMMARY:
Phase I/II trial to study the effectiveness of combining yttrium Y 90 ibritumomab tiuxetan with rituximab in treating patients who have localized or recurrent lymphoproliferative disorder after an organ transplant. Monoclonal antibodies such as yttrium Y 90 ibritumomab tiuxetan and rituximab can locate cancer cells and either kill them or deliver radioactive cancer-killing substances to them without harming normal cells

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the safety and tolerability of yttrium Y 90 ibritumomab tiuxetan (IDEC-Y2B8) in patients with post-transplant lymphoproliferative disorder.

II. Determine the safety and toxicity profile of IDEC-Y2B8 and rituximab in these patients.

III. Correlate the Epstein-Barr virus viral load with response and relapse in patients treated with this regimen.

OUTLINE: This is a multicenter, dose-escalation study of yttrium Y 90 ibritumomab tiuxetan (IDEC-Y2B8).

Phase I: Patients receive rituximab IV and indium In 111 ibritumomab tiuxetan IV over 10 minutes on day 1. Patients undergo 2 (or 3 if needed) imaging scans between days 1-6. In the absence of altered biodistribution, patients receive rituximab IV followed within 4 hours by IDEC-Y2B8 IV over 10 minutes on day 8.Cohorts of 6 patients receive escalating doses of IDEC-Y2B8 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which no more than 1 of 6 patients experience dose-limiting toxicity.

Phase II: Patients receive treatment as in phase I at the MTD of IDEC-Y2B8. Patients are followed monthly for 3 months, every 3 months for 2 years, and then every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed post-transplant lymphoproliferative disorder (PTLD) of 1 of the following stages:

  * Stage III or IV
  * Localized (not amenable to localized radiotherapy or excision)
  * Recurrent
* The following histologies* are eligible:

  * Polyclonal PTLD
  * Monoclonal PTLD
  * Diffuse large B-cell non-Hodgkin's lymphoma (NHL)
  * Lymphoplasmacytic NHL
  * Burkitt/Burkitt-like NHL
* Must not have completely responded during OR progressed after prior rituximab with or without chemotherapy

  * No history of rapid disease progression while receiving prior chemotherapy
* Measurable disease
* Must have less than 25% bone marrow involvement with lymphoma
* Prior solid organ transplantation required
* Evaluation of malignant cells for Epstein-Barr virus (EBV) required

  * EBV positive or negative allowed
* No pleural effusion
* No CNS lymphoma, including leptomeningeal disease
* No pulmonary involvement by NHL in patients with prior lung transplantation
* No HIV or AIDS-related lymphoma
* No hypocellular bone marrow (i.e., less than 15% cellularity)
* No marked reduction in bone marrow precursors of one or more cell lines (i.e., granulocytic, megakaryocytic, or erythroid)
* Performance status - Karnofsky 50-100%
* At least 3 months
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 150,000/mm^3
* Bilirubin no greater than 2.5 mg/dL
* Creatinine no greater than 2.5 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after study participation
* HIV negative
* No serious nonmalignant disease or infection that would compromise study objectives
* No presence of antimurine antibody reactivity
* No other concurrent active malignancy requiring therapy
* More than 2 weeks since prior filgrastim (G-CSF) or sargramostim (GM-CSF)
* More than 6 weeks since prior rituximab
* No prior allogeneic bone marrow or hematopoietic stem cell transplantation
* No prior radioimmunotherapy for NHL
* More than 4 weeks since prior chemotherapy
* See Biologic therapy
* No prior radiotherapy to more than 25% of active bone marrow (involved field or regional)
* More than 4 weeks since prior major surgery except diagnostic surgery
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2003-07; Primary Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Response rate | Up to 4 years
  Estimated using binomial proportions and their 95% confidence intervals.

SECONDARY OUTCOMES:
Time to response | Up to 4 years
  Analyzed by the Kaplan-Meier non-parametric methods.
Time to progression | From the date of first study treatment to the first date when progressive disease is documented, assessed up to 4 years
  Analyzed by the Kaplan-Meier non-parametric methods.
Incidence of toxicity related dose reductions graded according to the NCI CTCAE version 3.0 | Up to 4 years
  Presented by severity for each dose group.

CONTACTS AND LOCATIONS:
Overall Officials: David Scadden, Principal Investigator — AIDS Associated Malignancies Clinical Trials Consortium
Locations (1):
- AIDS - Associated Malignancies Clinical Trials Consortium, Rockville, Maryland, United States